CLINICAL TRIAL: NCT04494646
Title: BARCONA: A Phase II, Randomized, Double-blind, Placebo-controlled, Multi-center Study of the Effects of Bardoxolone Methyl in Participants With SARS-Corona Virus-2 (COVID-19)
Brief Title: BARCONA: A Study of Effects of Bardoxolone Methyl in Participants With SARS-Corona Virus-2 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Reata Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-00591
Record Dates: First submitted 2020-07-29; First posted 2020-07-31 (Actual); Results first posted 2022-01-12 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: Bardoxolone Methyl
MeSH Terms: conditions — COVID-19 | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All patients, investigators, site personnel, laboratories, and study personnel with direct involvement in the conduct of the study or their designees will be blinded to treatment assignments. To prevent potential bias, appropriate measures will be taken to ensure the blind is maintained for the patients and personnel mentioned previously. To maintain the blind, investigators will distribute blinded study drug treatment to patients as directed by the IWRS system. Investigators and patients will not be blinded to dose level, but will be blinded to treatment assignment (i.e., bardoxolone methyl vs. placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bardoxolone Methyl (Experimental): Patients will be randomized using permuted block randomization in a 1:1 fashion to either once-daily administration of bardoxolone methyl (20 mg) or matching placebo
  Interventions: Drug: Bardoxolone Methyl
- Placebo (Placebo Comparator): Patients will be randomized using permuted block randomization in a 1:1 fashion to either once-daily administration of bardoxolone methyl (20 mg) or matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bardoxolone Methyl — Once-daily administration of bardoxolone methyl (20mg)
  Arms: Bardoxolone Methyl
Drug: Placebo — Once-daily administration of matching placebo
  Arms: Placebo

SUMMARY:
This multi-center, double-blind, placebo-controlled, randomized Phase 2 trial will study the safety, tolerability, and efficacy of bardoxolone methyl in patients hospitalized with confirmed COVID-19. The trial will include approximately 40 patients and is designed to provide an early interim analysis of safety. Patients will be randomized using permuted block randomization in a 1:1 fashion to either once-daily administration of bardoxolone methyl (20 mg) or matching placebo and treatment will be administered for the duration of hospitalization (until recovery), with a maximum treatment duration of 29 days.

DETAILED DESCRIPTION:
Following randomization on Day 1, patients will be assessed while hospitalized on Days 3, 5, 8, 11, 15, 22, and 29. Assessments will include clinical status assessments, vital sign measurements, clinical chemistry collection, and adverse event collection. Patients that recover prior to Day 29 will complete an end-of-treatment visit. Patients will have an in-person follow-up on Day 29, regardless of treatment adherence and recovery status prior to Day 29, and a safety follow-up 60 days after randomization for clinical status assessments, vital sign measurements, clinical chemistry collection, and adverse event collection. Follow-up in-person visits are preferred but recognizing quarantine and other factors may limit the subject's ability to return to the site for the visit. In this case, the visit may be performed by phone. An independent Data and Safety Monitoring Board will advise the study leadership on safety aspects and overall progress of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Laboratory-confirmed COVID-19 infection as determined by polymerase chain reaction (PCR)
2. Hospitalized patients that meets one of the following conditions:

   1. Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.); OR
   2. At rest, blood oxygen saturation ≤ 94%; OR
   3. Require supplemental oxygen; OR
   4. Requiring non-invasive ventilation; OR
   5. Requiring invasive mechanical ventilation for up to 2 days.
3. Age ≥ 18 years. Enrollment of patients ≥70 years of age may be limited (e.g., comprise no more than 10% of all randomized patients), pending safety review by the DSMB and executive committee
4. Participant or legally authorized representative is willing to give informed consent

Exclusion Criteria:

1. Intubated and on invasive mechanical ventilation for three or more days at the time of randomization
2. Known left ventricular ejection fraction (LVEF) <40% or prior hospitalization for heart failure
3. Cardiac arrest
4. Shock
5. Known uncontrolled bacterial, fungal, or non-COVID viral infection
6. eGFR <30 ml/min/1.73 m² or requiring dialysis
7. ALT or AST > 5X ULN
8. History of cirrhosis, chronic active hepatitis or severe hepatic disease
9. Pregnant or lactating women
10. Enrolled in other trial of unapproved therapies, unless approved by trial Principal Investigator. In general, co-enrollment will be permitted unless there are safety concerns, mechanistic incompatibility or inability to adjudicate serious adverse events and will be decided on a case by case basis.
11. If in the opinion of the clinical team, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sripal Bangalore, MD, MHA, Principal Investigator — NYU Langone Health
Locations (8):
- United States (8):
  - HSHS St. John's Hospital (Prairie Education and Research Cooperative), Springfield, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - Coney Island Hospital, Brooklyn, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - NYU Winthrop Hospital, Mineola, New York
  - NYU Bellevue Hospital Center, New York, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Sripal.Bangalore@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bardoxolone Methyl | Placebo
Started | 21 | 19
Completed | 21 | 17
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bardoxolone Methyl | Placebo | Total
Number analyzed (Participants) | 21 | 17 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (16.3) | 60.5 (12.5) | 57.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 16 | 11 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 16 | 9 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events
Time Frame: Day 29
Measure: Number; unit: Adverse Events
Arm/Group | Bardoxolone Methyl | Placebo
Number analyzed (Participants) | 21 | 17
Adverse Events | 4 | 6

ADVERSE EVENTS:
Time Frame: 29 Days
Arm/Group | Bardoxolone Methyl | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 4/17
Serious Adverse Events (participants affected / at risk) | 4/21 | 6/17
Other Adverse Events (participants affected / at risk) | 1/21 | 1/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bardoxolone Methyl (N=21) | Placebo (N=17)
Presyncope, Pre-syncope (Nervous system disorders) | 0 | 1
Hypoxia, Worsening hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardiac failure acute, Acute on chronic systolic (congestive) heart failure (Cardiac disorders) | 0 | 1
Nephrolithiasis, Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Mechanical ventilation, Invasive mechanical ventilation (Surgical and medical procedures) | 1 | 0
Abdominal wall wound, Worsening abdominal wound (Injury, poisoning and procedural complications) | 1 | 0
Respiratory failure Worsening hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mechanical ventilation (Surgical and medical procedures) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Pneumonia due to covid-19 virus (Infections and infestations) | 1 | 0
Splenic laceration (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bardoxolone Methyl (N=21) | Placebo (N=17)
Dizziness and Lightheadedness (Nervous system disorders) | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 1 | 0
Blackouts (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04494646/Prot_SAP_000.pdf